CLINICAL TRIAL: NCT03067181
Title: A Phase 3 Study of Active Surveillance for Low Risk and a Randomized Trial of Carboplatin vs. Cisplatin for Standard Risk Pediatric and Adult Patients With Germ Cell Tumors
Brief Title: Active Surveillance, Bleomycin, Etoposide, Carboplatin or Cisplatin in Treating Pediatric and Adult Patients With Germ Cell Tumors
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGCT1531; NCI-2017-00178 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AGCT1531; AGCT1531 (Other: Children's Oncology Group); AGCT1531 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2017-02-14; First posted 2017-03-01 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-06

CONDITIONS: Childhood Extracranial Germ Cell Tumor; Extragonadal Embryonal Carcinoma; Germ Cell Tumor; Malignant Germ Cell Tumor; Malignant Ovarian Teratoma; Stage I Ovarian Choriocarcinoma; Stage I Ovarian Embryonal Carcinoma AJCC v6 and v7; Stage I Ovarian Yolk Sac Tumor AJCC v6 and v7; Stage I Testicular Choriocarcinoma AJCC v6 and v7; Stage I Testicular Embryonal Carcinoma AJCC v6 and v7; Stage I Testicular Seminoma AJCC v6 and v7; Stage I Testicular Yolk Sac Tumor AJCC v6 and v7; Stage II Ovarian Choriocarcinoma; Stage II Ovarian Embryonal Carcinoma AJCC v6 and v7; Stage II Ovarian Yolk Sac Tumor AJCC v6 and v7; Stage II Testicular Choriocarcinoma AJCC v6 and v7; Stage II Testicular Embryonal Carcinoma AJCC v6 and v7; Stage II Testicular Yolk Sac Tumor AJCC v6 and v7; Stage III Ovarian Choriocarcinoma; Stage III Ovarian Embryonal Carcinoma AJCC v6 and v7; Stage III Ovarian Yolk Sac Tumor AJCC v6 and v7; Stage III Testicular Choriocarcinoma AJCC v6 and v7; Stage III Testicular Embryonal Carcinoma AJCC v6 and v7; Stage III Testicular Yolk Sac Tumor AJCC v6 and v7; Stage IV Ovarian Choriocarcinoma; Stage IV Ovarian Embryonal Carcinoma AJCC v6 and v7; Stage IV Ovarian Yolk Sac Tumor AJCC v6 and v7; Testicular Mixed Choriocarcinoma and Embryonal Carcinoma; Testicular Mixed Choriocarcinoma and Teratoma; Testicular Mixed Choriocarcinoma and Yolk Sac Tumor
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Carcinoma, Embryonal; Teratoma; Endodermal Sinus Tumor | interventions — Practice Guidelines as Topic; Standard of Care; Biopsy; Specimen Handling; Bleomycin; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Etoposide; Magnetic Resonance Spectroscopy; Pharmacogenomic Testing; Respiratory Physiological Phenomena

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm I (bleomycin, carboplatin, etoposide) (Experimental): Patients receive bleomycin IV over 10 minutes and carboplatin IV over 1 hour on day 1. Patients also receive etoposide IV over 1-2 hours on days 1-5. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT, MRI, and/or chest x-ray as well as blood sample collection throughout the trial. Patients may also undergo a tumor biopsy throughout the trial. Patients undergo a pulmonary function test on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Biological: Bleomycin Sulfate; Drug: Carboplatin; Procedure: Computed Tomography; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Other: Pharmacogenomic Study; Procedure: Pulmonary Function Test; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (bleomycin, etoposide, cisplatin) (Experimental): Patients receive bleomycin IV over 10 minutes on day 1. Patients also receive etoposide IV over 1-2 hours and cisplatin IV over 1-3 hours on days 1-5. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT, MRI, and/or chest x-ray as well as blood sample collection throughout the trial. Patients may also undergo a tumor biopsy throughout the trial. Patients undergo a pulmonary function test on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Biological: Bleomycin Sulfate; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Other: Pharmacogenomic Study; Procedure: Pulmonary Function Test; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm III (bleomycin, etoposide, carboplatin) (Experimental): Patients receive bleomycin IV over 10 minutes on days 1, 8, and 15, etoposide IV over 1-2 hours on days 1-5, and carboplatin IV over 1 hour on day 1. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT, MRI, and/or chest x-ray as well as blood sample collection throughout the trial. Patients may also undergo a tumor biopsy throughout the trial. Patients undergo a pulmonary function test on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Biological: Bleomycin Sulfate; Drug: Carboplatin; Procedure: Computed Tomography; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Other: Pharmacogenomic Study; Procedure: Pulmonary Function Test; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm IV (bleomycin, etoposide, cisplatin) (Experimental): Patients receive bleomycin IV over 10 minutes on days 1, 8, and 15, etoposide IV over 1-2 hours on days 1-5, and cisplatin IV over 1-3 hours on days 1-5. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT, MRI, and/or chest x-ray as well as blood sample collection throughout the trial. Patients may also undergo a tumor biopsy throughout the trial. Patients undergo a pulmonary function test on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Biological: Bleomycin Sulfate; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Other: Pharmacogenomic Study; Procedure: Pulmonary Function Test; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Low-Risk (observation) (Experimental): Patients with low-risk stage I grade 2, 3 ovarian immature teratoma or stage I non-seminoma or seminoma MGCTs undergo observation and can transfer to standard risk arm when eligibility criteria are met. Patients with stage I seminoma testicular MGCT undergo observation, and those with residual/recurrent disease are treated at the discretion of their physician. Patients undergo CT, MRI, and/or chest x-ray as well as blood sample collection throughout the trial. Patients may also undergo a tumor biopsy throughout the trial.
  Interventions: Other: Best Practice; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Pharmacogenomic Study; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Undergo observation
  Other Names: standard of care; standard therapy
  Arms: Low-Risk (observation)
Procedure: Biopsy Procedure — Undergo a tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Bleomycin Sulfate — Given IV
  Other Names: Blanoxan; BleMomycine; Blenoxane; Bleo-cell; Bleo-S; Bleocin; Bleolem; Bleomycin Sulfas; Bleomycin Sulphate; Bleomycini Sulfas; Blexane; Oil Bleo
  Arms: Arm I (bleomycin, carboplatin, etoposide); Arm II (bleomycin, etoposide, cisplatin); Arm III (bleomycin, etoposide, carboplatin); Arm IV (bleomycin, etoposide, cisplatin)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm I (bleomycin, carboplatin, etoposide); Arm III (bleomycin, etoposide, carboplatin)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm II (bleomycin, etoposide, cisplatin); Arm IV (bleomycin, etoposide, cisplatin)
Procedure: Computed Tomography — Undergo a CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
  Arms: Arm I (bleomycin, carboplatin, etoposide); Arm II (bleomycin, etoposide, cisplatin); Arm III (bleomycin, etoposide, carboplatin); Arm IV (bleomycin, etoposide, cisplatin)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Pharmacogenomic Study — Correlative studies
  Other Names: PHARMACOGENOMIC
Procedure: Pulmonary Function Test — Undergo a pulmonary function test
  Other Names: lung function test; PFT; Pulmonary Function Testing; Pulmonary Function Tests
  Arms: Arm I (bleomycin, carboplatin, etoposide); Arm II (bleomycin, etoposide, cisplatin); Arm III (bleomycin, etoposide, carboplatin); Arm IV (bleomycin, etoposide, cisplatin)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial studies how well active surveillance help doctors to monitor subjects with low risk germ cell tumors for recurrence after their tumor is removed. When the germ cell tumor has spread outside of the organ in which it developed, it is considered metastatic. Chemotherapy drugs, such as bleomycin, carboplatin, etoposide, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. The trial studies whether carboplatin or cisplatin is the preferred chemotherapy to use in treating metastatic standard risk germ cell tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether a strategy of complete surgical resection followed by surveillance can maintain an overall survival rate of at least 95.7% at two years for pediatric, adolescent and adult patients with stage I (low risk) malignant germ cell tumors (Stratum 2), and at least 88% for patients with all stage/grade ovarian pure immature teratoma (Stratum 1).

II. To compare the event-free survival of a carboplatin versus (vs.) cisplatin-based regimen in the treatment of pediatric, adolescent and young adult patients with standard risk non-seminomatous germ cell tumors.

IIa. To compare the event free survival (EFS) of a carboplatin-based regimen (carboplatin [C] etoposide [E] bleomycin [b]) vs. a cisplatin-based regimen (cisplatin [P]Eb) in children (less than 11 years in age) with standard risk germ cell tumors (GCT).

IIb. To compare the EFS of a carboplatin-based regimen (BEC) vs. a cisplatin-based regimen (BEP) in adolescents and young adults (ages 11 - < 25 years) with standard risk GCT.

SECONDARY OBJECTIVES:

I. To compare the incidence of ototoxicity in children, adolescents and young adults with standard risk germ cell tumors treated with carboplatin-based chemotherapy as compared to cisplatin-based chemotherapy.

II. To refine and validate a novel patient-reported measure of hearing outcomes for children, adolescents and young adults with standard risk germ cell tumors.

III. To determine whether radiomic measures of body composition at diagnosis, end of therapy, and one year after end of therapy is better correlated with adverse events compared to body surface area in patients receiving chemotherapy for germ cell tumors.

EXPLORATORY OBJECTIVES:

I. To prospectively determine the correlation of tumor marker decline (alpha-fetoprotein [FP] and beta-human chorionic gonadotropin [HCG]) with clinical outcome in low and standard risk germ cell tumor patients.

II. To compare self-reported peripheral neuropathy and other patient-reported outcomes between children, adolescents and young adults with standard risk germ cell tumors treated with carboplatin-based chemotherapy as compared to cisplatin-based chemotherapy.

III. Assess the relationship between hearing loss as measured by audiometry with the effects of tinnitus as assessed on the Adolescent and Young Adult Hearing Screening (AYA-HEARS) instrument.

IV. To evaluate the prognostic significance of serum micro ribonucleic acid (miRNA)s in stage I testicular cancer (seminoma and non-seminoma) patients by collecting clinical data and serum specimens for future analysis.

V. To compare differences in the proportion of patients with residual mass(es) ≥ 1 cm at the completion of chemotherapy among patients randomized to the cisplatin and carboplatin-containing arms and to compare the proportion undergoing post-chemotherapy surgery for residual mass(es), and the proportion of resected masses with viable malignancy, teratoma, or necrosis.

OUTLINE:

Patients with low-risk stage I grade 2, 3 ovarian immature teratoma or stage I non-seminoma malignant germ cell tumors (MGCT)s undergo observation and can transfer to standard risk arm at time of recurrence if eligibility criteria are met. Patients with stage I seminoma testicular MGCT undergo observation, and those with residual/recurrent disease are treated at the discretion of their physician. Patients undergo computed tomography (CT), magnetic resonance imaging (MRI), and/or chest x-ray as well as blood sample collection throughout the trial to monitor for response and recurrence. Patients may also undergo a tumor biopsy throughout the trial.

Patients with standard risk 1 are randomized into 1 of 2 arms.

ARM I (CEb): Patients receive bleomycin intravenously (IV) over 10 minutes and carboplatin IV over 1 hour on day 1. Patients also receive etoposide IV over 1-2 hours on days 1-5. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT, MRI, and/or chest x-ray as well as blood sample collection throughout the trial. Patients may also undergo a tumor biopsy throughout the trial. Patients undergo a pulmonary function test on study.

ARM II (PEb): Patients receive bleomycin IV over 10 minutes on day 1. Patients also receive etoposide IV over 1-2 hours and cisplatin IV over 1-3 hours on days 1-5. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT, MRI, and/or chest x-ray as well as blood sample collection throughout the trial. Patients may also undergo a tumor biopsy throughout the trial. Patients undergo a pulmonary function test on study.

Patients with standard risk 2 are randomized into 1 of 2 arms.

ARM III (BEC): Patients receive bleomycin IV over 10 minutes on days 1, 8, and 15, etoposide IV over 1-2 hours on days 1-5, and carboplatin IV over 1 hour on day 1. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT, MRI, and/or chest x-ray as well as blood sample collection throughout the trial. Patients may also undergo a tumor biopsy throughout the trial. Patients undergo a pulmonary function test on study.

ARM IV (BEP): Patients receive bleomycin IV over 10 minutes on days 1, 8, and 15, etoposide IV over 1-2 hours on days 1-5, and cisplatin IV over 1-3 hours on days 1-5. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT, MRI, and/or chest x-ray as well as blood sample collection throughout the trial. Patients may also undergo a tumor biopsy throughout the trial. Patients undergo a pulmonary function test on study.

After completion of study treatment, patients are followed up every 2 months for 12 months, every 3-6 months to 24 months, every 6 months for years 3-5, and then annually for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* There is no age limit for the low risk stratum (stage I ovarian immature teratoma and stage I non-seminoma or seminoma malignant GCT [all sites])
* Standard risk 1: Patients must be < 11 years of age at enrollment
* Standard risk 2: Patients must be >= 11 and < 25 years of age at enrollment
* Patients enrolling on one of the low risk arms must be newly diagnosed with a stage I germ cell tumor; for the standard risk arms, patients must be newly diagnosed with malignant germ cell tumor (stage II or higher).

  * Histologic confirmation of a primary extracranial germ cell tumor in any of the categories outlined below is required of all patients at enrollment , with the following exceptions:

    * Among patients were initially diagnosed with completely resected non-seminoma malignant GCT and later recur during observation post surgery, a diagnostic biopsy is not required for enrollment if elevated tumor markers rise to > 5 x upper limit of normal (ULN) on at least 2 measurements taken at least 1 week apart. The pathology report of initial surgery should be provided
    * Patients may be enrolled without histologic or cytologic confirmation in the rare case where there are exceptionally raised tumor markers (alpha fetoprotein [AFP- ≥ 500 ng/mL or HCG ≥ 500 IU/L) and radiologic features consistent with GCT. In addition, the treating clinician must deem that the patient's tumor is not suitable for upfront resection and that a biopsy is not in the patient's best interest; or that there is a need to start therapy urgently
* Low risk immature teratoma (IT); site: ovarian; stage: any; grade: any; histology: pure immature teratoma, mixed immature and mature teratoma, (may contain microscopic foci of yolk sac tumor [< 3 mm], but no other pathological evidence of MGCT); tumor markers: alpha-FP =< 1,000 ng/mL, beta-HCG institutional normal; all ages
* Low risk stage I non-seminoma MGCT; site: ovarian, testicular, or extragonadal; stage: COG stage I, FIGO stage IA and IB, American Joint Committee on Cancer (AJCC) testicular stage IA, IB and IS; histology: must contain at least one of the following: yolk sac tumor, embryonal carcinoma, or choriocarcinoma (pure or mixed); all ages
* Low risk stage I seminoma-MGCT; site: testicular; stage: COG stage I; AJCC testicular stage IA IB, and IS; histology: must contain only seminoma; may contain immature/mature teratoma; may NOT contain yolk sac tumor, embryonal carcinoma, or choriocarcinoma; all ages
* Standard risk 1 (SR1); site: ovarian, testicular, or extragonadal; stage: COG stage II-IV, FIGO stage IC-IV, (International Germ Cell Consensus Classification [IGCCC] criteria DO NOT apply); histology: must contain at least one of the following: yolk sac tumor, embryonal carcinoma, or choriocarcinoma; age (years) < 11
* Standard risk 2 (SR2)

  * Site: ovarian; stage: COG stage II, III, and III-X, FIGO stage IC, II and III; histology: must contain at least one of the following: yolk sac tumor, embryonal carcinoma, or choriocarcinoma; age (years) >= 11 and < 25
  * Site: testicular; stage: COG stage II-IV, AJCC stage II, III, IGCCC good risk; histology: must contain at least one of the following: yolk sac tumor, embryonal carcinoma, or choriocarcinoma: must be IGCCC good risk; post op: alpha-FP < 1,000 ng/mL, beta-HCG < 5,000 IU/mL and lactate dehydrogenase (LDH) < 3.0 x normal; age (years) >= 11 and < 25
* Notes:

  * IGCCC criteria only apply to SR2 patients with a testicular primary tumor
  * Use post-op tumor marker levels to determine IGCCC risk group
  * Pure seminoma patients are not eligible for the standard risk arms of the study
  * For the low risk stage I non-seminoma MGCT and the standard risk arms, components of yolk sac tumor, embryonal carcinoma, or choriocarcinoma can be mixed with other forms of GCT, such as seminoma or mature or immature teratoma; if yolk sac tumor is the only malignant component present, then it must be deemed by the pathologist to be greater than a "microscopic component" of yolk sac tumor
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, 2 or 3; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Organ function requirements apply ONLY to patients who will receive chemotherapy (SR1 and SR2 patients)
* Adequate renal function defined as:
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 (within 7 days prior to enrollment) OR
* A serum creatinine based on age/sex as follows (within 7 days prior to enrollment): (mg/dL)

  * 1 month to < 6 months male: 0.4 female: 0.4
  * 6 months to < 1 year male: 0.5 female: 0.5
  * 1 to < 2 years male: 0.6 female: 0.6
  * 2 to < 6 years male: 0.8 female: 0.8
  * 6 to < 10 years male: 1 female: 1
  * 10 to < 13 years male: 1.2 female: 1.2
  * 13 to < 16 years: male: 1.5 female: 1.4
  * >= 16 years male: 1.7 female: 1.4
* Total bilirubin =< 2 x upper limit of normal (ULN) for age (within 7 days prior to enrollment)

  * Unless due to Gilbert's disease, malignant involvement of liver or vanishing bile duct syndrome
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x upper limit of normal (ULN) (within 7 days prior to enrollment)

  * Unless due to Gilbert's disease, malignant involvement of liver or vanishing bile duct syndrome
* Peripheral absolute neutrophil count (ANC) >= 750/mm^3 (within 7 days prior to enrollment) AND
* Platelet count >= 75,000/mm^3 (within 7 days prior to enrollment)
* Patients enrolling on the standard risk arms must be medically fit to receive protocol treatment and with no contraindications to protocol treatment
* Eligibility criteria to participate in the pilot study of the AYA-Hears instrument (patient reported outcomes [PROs] of ototoxicity) Note: participants in group 1 will not receive AGCT1531 protocol-directed therapy; all other AYA-HEARS patients must be enrolled on the AGCT1531 SR2 arm in order to participate
* >= 11 and < 25 years old at enrollment
* Able to fluently speak and read English
* Has received prior cisplatin- or carboplatin-based chemotherapy regimen for malignancy including diagnoses other than germ cell tumor
* Followed for cancer or survivorship care at one of the following institutions:

  * Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center
  * Dana Farber/Harvard Cancer Center
  * Hospital for Sick Children
  * Children's Hospital of Eastern Ontario
  * Oregon Health and Science University
  * Seattle Children's Hospital
  * Yale University

Exclusion Criteria:

* Patients with any diagnoses not listed including:

  * Stage I testicular cancer patients who have undergone primary RPLND (retroperitoneal lymph node dissection)
  * Pure ovarian or extragonadal dysgerminoma/seminoma
  * Pure mature teratoma
  * Pure immature teratoma with alpha-fetoprotein (AFP) >= 1000 ng/mL
  * "Poor risk" GCT (age >= 11 years old and COG stage IV ovarian, COG stage II- IV extragonadal, or IGCCC intermediate or poor risk testicular), or
  * Primary central nervous system (CNS) germ cell tumor
  * Germ cell tumor with somatic malignant transformation
  * Spermatocytic seminoma
* Patients must have had no prior systemic therapy for the current cancer diagnosis
* Patients must have had no prior radiation therapy with the exception of CNS irradiation of brain metastases; (this exception only applies to SR1 patients; any patients over age 11 with distant metastases to brain [stage IV disease] would be considered poor risk and therefore not eligible for this trial)
* Patients with significant, pre-existing co-morbid respiratory disease that contraindicate the use of bleomycin are ineligible for the standard risk arms of the trial
* Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs; a pregnancy test is required for female patients of childbearing potential; (this criteria applies ONLY to patients who will receive chemotherapy [SR1 and SR2 patients])
* Lactating females who plan to breastfeed their infants; (this criteria applies ONLY to patients who will receive chemotherapy [SR1 and SR2 patients])
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation; (this criteria applies ONLY to patients who will receive chemotherapy [SR1 and SR2 patients])

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1780 (Estimated)
Dates: Start 2017-05-25 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Two years post enrollment
  The time from study entry to the date of death, or date of last contact and ascertained as alive, whichever comes first.
Event-free survival | Two years post enrollment
  The time from study entry to the date of death, date of disease progression or recurrence, date of second malignant neoplasm or date of last contact and ascertained as alive, whichever comes first.

SECONDARY OUTCOMES:
Proportion of participants with hearing loss | 8 weeks after the last dose of platin therapy
  The hearing loss is evaluated according to the International Society of Pediatric Oncology criteria.
Number of participants by understanding score category in the Adolescents and Young Adults-Hearing Screen | Baseline
  Understanding score will be rated on a 5-point Likert scale ranging from 0 = completely incorrect to 4 = completely correct.
Correlation of radiomic measures of body composition to ototoxicity, neurotoxicity, or hematologic toxicity compared to body surface area | At diagnosis, at end of therapy, and up to 1 year after end of therapy
  Imaging and radiology reports will be analyzed using Slice-O-Matic software (Tomovision), and imaging results will be used to calculate whole-body lean body mass. Will fit logistic regression models to quantify the association between dose defined by body composition and the presence of toxicity (ototoxicities, neurotoxicities, and hematologic toxicities).

OTHER OUTCOMES:
Event-free survival (EFS) for participants with and without tumor marker decline | Up to 2 years
  Tumor marker decline is coded as yes versus no. The hazard ratio for participants with and without tumor marker decline will be presented. Patients who receive chemotherapy will be analyzed separately than patients in the low risk stratum.
Mean self-reported peripheral neuropathy score | Up to 12 months
  Mean self-reported neuropathy score will be compared for the two treatment regimens.
Differences in the proportion of patients with residual mass(es) ≥ 1 cm | Up to 12 months
  Will conduct a 2-sample test of proportions to compare the proportion of patients with residual tumors at the completion of therapy between the cisplatin and carboplatin arms stratified by age group (SR1 and SR2). Will use a significance level of 0.05 to test the null hypothesis that the proportion of patients with residual tumor at the end of therapy is the same for both treatment arms.Will compare the proportion of patients undergoing post-chemotherapy surgery for residual masses. Will describe the proportion of patients with viable malignancy, teratoma, or necrosis. Will describe the above proportions by tumor site (testicular, ovarian, and extra gonadal). If imaging reports are missing for a large proportion of patients, will also fit logistic regression models to compare the odds of residual tumor after adjusting for potential confounders. Separate models will be fit for SR1 and SR2 patients.

CONTACTS AND LOCATIONS:
Overall Officials: A. L Frazier, Principal Investigator — Children's Oncology Group
Locations (629):
- United States (566):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Banner Children's at Desert, Mesa, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Kaiser Permanente-Fontana, Fontana, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Providence Queen of The Valley, Napa, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Woodland Memorial Hospital, Woodland, California
  - Children's Hospital Colorado, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - UCHealth Lone Tree Health Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Saint John's Hospital, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Blank Children's Hospital, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - The Iowa Clinic PC, West Des Moines, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Cancer Care Specialists - Reno, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Glens Falls Hospital, Glens Falls, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Westchester Medical Center, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Novant Health Cancer Institute - Rowan, Salisbury, North Carolina
  - Rowan Regional Medical Center, Salisbury, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - OhioHealth O'Bleness Hospital, Athens, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Memorial Hospital, Marysville, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - OhioHealth Pickerington Methodist Hospital, Pickerington, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - OhioHealth Westerville Medical Campus/Westerville Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - North Grove Medical Park, Spartanburg, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Spartanburg Medical Center - Mary Black Campus, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Texas Tech University Health Sciences Center-El Paso, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
- Australia (8):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Monash Medical Center-Clayton Campus, Clayton, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- Canada (17):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- Tata Memorial Hospital, Mumbai, India
- Japan (17):
  - Tohoku University School of Medicine, Sendai, Aoba-ku
  - Chiba University, Chiba-sgi, Chiba
  - Niigata Cancer Centre, Niigata, Chuo-ku
  - Kyushu Univeristy, Higashiku, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Prefectural Kobe Children's Hospital, Kobe, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Kanagawa Children's Medical Center, Yokohama, Kanagawa
  - Saitama Children's Medical Center, Chuo-ku, Saitama
  - Keio University, Shinjuku-ku, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - Kyoto Perfectural University of Medicine, Kyoto
  - Hyogo College of Medicine, Nishinomiya, Hyogo
  - Osaka City General Hospital, Osaka
  - Saitama Medical University International Medical Center, Saitama
  - National Cancer Center Hospital, Tokyo
  - Kokuritsu Seiiku Medical Research Center Hospital, Tokyo
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- Puerto Rico (2):
  - HIMA San Pablo Oncologic Hospital, Caguas
  - San Jorge Children's Hospital, San Juan
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia
- United Kingdom (15):
  - Sheffield Children's Hospital, Broomhall, England
  - Addenbrookes Hospital-Medical School, Cambridge, England
  - Saint Bartholomew's Hospital, London, England
  - University College London Hospitals NHS Trust - Foley Street, London, England
  - Royal Manchester Children Hospital, Manchester, England
  - Royal Victoria Infirmary, Newcastle, England
  - Freeman Hospital, Newcastle upon Tyne, England
  - John Radcliffe Hospital, Oxford, England
  - Weston Park Hospital, Sheffield, England
  - Saint James's University Hospital, West Yorkshire, England
  - Western General Hospital, Edinburgh, Scotland
  - Royal Hospital for Children and Young People, Edinburgh, Scotland
  - Beatson Oncology Center, Glasgow, Scotland
  - Royal Hospital for Children, Glasgow, Scotland
  - Leeds General Infirmary, West Yorkshire

REFERENCES:
- [Derived] Trozzi R, Rosati A, Panico C, Perisiano C, Santoro A, Fagotti A. Extra-cranial meningioma associated with relapse of immature ovarian teratoma. Int J Gynecol Cancer. 2023 Oct 2;33(10):1649-1654. doi: 10.1136/ijgc-2023-004718. No abstract available. PMID 37783480